CLINICAL TRIAL: NCT03750383
Title: A Non-Randomized, Open-Label, Two-Part, Drug-Drug Interaction Study to Evaluate the Effects of Cyclosporine and Prednisone on the Pharmacokinetics and Safety of EDP-938 in Healthy Adult Subjects
Brief Title: Drug-Drug Interaction Study Between EDP-938, Cyclosporine and Prednisone in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Collaborators: Pharmaceutical Research Associates (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EDP 938-002
Record Dates: First submitted 2018-11-08; First posted 2018-11-23 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2018-10

CONDITIONS: RSV Infection
Keywords: drug drug interaction study
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — EDP-938; Cyclosporine; Prednisone

STUDY DESIGN:
Intervention Model Description: 2-Part Single Group study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EDP-938 and cyclosporine interaction (Part 1) (Experimental)
  Interventions: Drug: EDP-938; Drug: Cyclosporine
- EDP-938 and prednisone interaction (Part 2) (Experimental)
  Interventions: Drug: EDP-938; Drug: Prednisone

INTERVENTIONS:
Drug: EDP-938 — Subjects will receive EDP-938 once daily on Day 1 and Day 5 (Part 1)
  Arms: EDP-938 and cyclosporine interaction (Part 1)
Drug: EDP-938 — Subjects will receive one dose of EDP-938 on Day 1 and Day 8 (Part 2)
  Arms: EDP-938 and prednisone interaction (Part 2)
Drug: Cyclosporine — Subjects will receive one dose of cyclosporine on Day 5
  Arms: EDP-938 and cyclosporine interaction (Part 1)
Drug: Prednisone — Subjects will receive prednisone once daily from Day 5 to Day 14
  Arms: EDP-938 and prednisone interaction (Part 2)

SUMMARY:
A Non-Randomized, Open-Label, Two-Part, Drug-Drug Interaction Study to Evaluate the Effects of Cyclosporine and Prednisone on the Pharmacokinetics and Safety of EDP-938 in Healthy Adult Subjects

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document signed and dated by the subject.
* Healthy male and female subjects of any ethnic origin between the ages of 18 and 55 years, inclusive.
* Screening body mass index (BMI) of 18 to 30 kg/m2 with a minimum body weight of 50 kg
* Female subjects of childbearing potential must agree to use two effective methods of contraception from the date of Screening until 90 days after the last dose of EDP 938.

Exclusion Criteria:

* Clinically relevant evidence or history of illness or disease.
* Pregnant or nursing females.
* History of febrile illness within 7 days prior to the first dose of study drug or subjects with evidence of active infection.
* A positive urine drug screen at screening or Day -1.
* Current tobacco smokers or use of tobacco within 3 months prior to screening.
* Any condition possibly affecting drug absorption (e.g., gastrectomy, cholecystectomy).
* History of regular alcohol consumption.
* Participation in a clinical trial within 30 days prior to the first dose of study drug.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2018-11-17 (Actual); Study Completion 2018-12-13 (Actual)

PRIMARY OUTCOMES:
Cmax of EDP-938 with and without coadministration with cyclosporine | Up to 12 days
AUC of EDP-938 with and without coadministration with cyclosporine | Up to 12 days
Cmax of EDP-938 with and without coadministration with prednisone | Up to 21 days
AUC of EDP-938 with and without coadministration with prednisone | Up to 21 days

SECONDARY OUTCOMES:
Safety measured by adverse events | Up to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Enanta Pharmaceuticals, Inc, Study Director — Enanta Pharmaceuticals, Inc
Locations (1):
- Pharmaceutical Research Associates, Inc.,, Lenexa, Kansas, United States